CLINICAL TRIAL: NCT06402578
Title: A Feasibility Randomised Controlled Trial to Investigate the Effects of a 12-week Digital Physical Activity Programme, With or Without Physical Education Support, on Blood Glucose Control in Patients With Type 2 Diabetes Mellitus
Brief Title: A 12-week Digital Physical Activity Programme, With or Without Physical Education Support for Type 2 Diabetes Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Phil Calvert, Principal Investigator, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: QMU-IRAS ID: 327162
Record Dates: First submitted 2024-03-13; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: HbA1c; Cholesterol; Resting Heart Rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: At the point of consent the participants will be randomised to one of three allocated groups. Control group, Intervention 1 or Intervention 2.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group, (No Intervention): Control Group, will be issued with a smartwatch that is paired with a freely accessible App called Alexia® to record their PA. They will be asked to carry on with their daily activity and to record when they do any of their own physical activities that they do themselves routinely on an everyday basis during the 12 week study. They will not receive a 12 week PA programme.
- Intervention 1 (Experimental): Intervention 1, will be provided with a 12 week PA programme and asked to record their PA while they follow the programme during the 12 week study.
  Interventions: Diagnostic Test: HbA1c testing
- Intervention 2 (Experimental): Intervention 2, will also be provided with the same 12 week PA program and asked to record their PA while they follow the programme during the 12 week study. The participants in this group will also get support from a physical activity professional (PAP) who will be monitoring their 12 week journey. The PAP will be prompting the participant with weekly information as to why they are doing these exercises as well as supporting the participants to continue their programme as soon as non-adherence to the exercise program becomes apparent during the 12 week study.
  Interventions: Diagnostic Test: HbA1c testing

INTERVENTIONS:
Diagnostic Test: HbA1c testing — Bloods will be take pre and post 12 week intervention.
  Arms: Intervention 1; Intervention 2

SUMMARY:
Investigation into the effects of a 12-week digital physical activity programme, with or without physical education support on blood glucose control in patients with T2DM using HbA1c testing.

DETAILED DESCRIPTION:
Primary objective: investigate the effects of a 12-week digital physical activity programme, with or without physical education support on blood glucose control in patients with T2DM using HbA1c testing. Secondary objective: evaluate the effects on Cholesterol (ratio of High Density Lipids to Low Density Lipids), Resting Heart Rate, and Body Mass Index after a 12 week physical activity programme. Monitor step counts and sleep patterns during a 12 week physical activity programme.: Methods: Using a RCT is intended to implement dependent variable inductive research into a 12-week e-Health Physical activity (PA) programme with or without physical education support focusing on the blood glucose control in patients with T2DM. Recruitment of 60 patients from hospital out-patient clinics, community diabetic departments, and. NHS patients from general practitioners.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of T2DM in the last 3 years.
* Age 18+ years.
* Uses the English language as a primary or secondary language with the ability to read and write.
* Lives in the United Kingdom.
* Has no medical reason preventing participation in regular physical activity.
* Has a SMART phone with access to the internet.

Exclusion Criteria:

* Physical inability to participate in 12 weeks of physical activity.
* Cardiac or cardiovascular surgery in the past 6 months.
* Musculoskeletal issues that could be aggravated whilst participating in regular physical activity.
* Presently participating in a weight loss programme.
* Unable to commit to the 12-week feasibility study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
HbA1c testing | 12 weeks
  blood will be take pre and post trial.

SECONDARY OUTCOMES:
Cholesterol ratio testing | 12 weeks
  blood will be take pre and post trial.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Calvert, MSc, Principal Investigator — PhD student
Locations (1):
- Queen Margret University Edinburgh, Edinburgh, Musselburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided